CLINICAL TRIAL: NCT00777790
Title: Antibody Responses to a Booster Dose of an Experimental Tetravalent (A, C, Y, and W-135) Meningococcal Diphtheria Toxoid Conjugate Vaccine, Menactra® in Adolescents Who Previously Received Menomune® or Menactra®
Brief Title: Study of a Booster Dose of Meningococcal Diphtheria Toxoid Conjugate Vaccine in Adolescents
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sanofi Pasteur, a Sanofi Company (Industry)
Responsible Party: Sponsor
Organization: Sanofi (Industry)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: MTA19
Record Dates: First submitted 2008-10-21; First posted 2008-10-22 (Estimated); Results first posted 2009-03-19 (Estimated); Last update posted 2014-02-14 (Estimated); Status verified 2014-01

CONDITIONS: Meningitis; Meningococcemia
Keywords: Meningitis; Meningococcemia; Neisseria meningitidis
MeSH Terms: conditions — Meningitis; Meningococcal Infections | interventions — Meningococcal Vaccines

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Menactra® Group (Experimental): Received Menactra® vaccine in Study MTA02
  Interventions: Biological: Meningococcal Polysaccharide Diphtheria Toxoid Conjugate
- Menomune® Group (Experimental): Received Menomune® vaccine in Study MTA02
  Interventions: Biological: Meningococcal Polysaccharide Diphtheria Toxoid Conjugate
- Control Group (Experimental): Meningococcal vaccine-naïve Control Group.
  Interventions: Biological: Meningococcal Polysaccharide Diphtheria Toxoid Conjugate

INTERVENTIONS:
Biological: Meningococcal Polysaccharide Diphtheria Toxoid Conjugate — 0.5 mL, Intramuscular
  Other Names: Menactra®
  Arms: Menactra® Group
Biological: Meningococcal Polysaccharide Diphtheria Toxoid Conjugate — 0.5 mL, Intramuscular
  Other Names: Menactra®
  Arms: Menomune® Group
Biological: Meningococcal Polysaccharide Diphtheria Toxoid Conjugate — 0.5 mL, Intramuscular
  Other Names: Mneactra®
  Arms: Control Group

SUMMARY:
This study was designed to evaluate the antibody response to a Menactra® booster dose in participants who previously received one dose of Menactra® or Menomune® as adolescents 3 years earlier in Study MTA02.

Primary Objective:

To evaluate the antibody responses to a booster dose of a tetravalent meningococcal diphtheria toxoid conjugate vaccine (Menactra®) in participants who had previously received Menactra® or Menomune® as adolescents in the MTA02 Study and antibody responses to a dose of Menactra® in naive adolescents.

DETAILED DESCRIPTION:
All subjects were given a single boosting dose of Menactra® to evaluate the kinetics of the response, the magnitude and the avidity of the antibody produced.

ELIGIBILITY:
Inclusion Criteria :

* Participant is healthy, as determined by medical history and physical examination.
* Participant is at least 13 years of age but not yet 22 years of age at time of enrollment.
* For the Menactra® and Menomune® groups, participant received one dose of Menactra® or Menomune® in MTA02 trial and completed trial (2 blood samples, contacted for Month 6 safety follow up).
* For the Control group, participant has no previous history of any meningococcal vaccination.
* If < 18 years of age, participant has signed Institutional Review Board (IRB) approved informed assent form and his/her parent/legal guardian has signed an IRB-approved informed consent form.
* If ≥ 18 years of age, participant has signed an IRB-approved informed consent form.
* Able to provide vaccination log.

Exclusion Criteria :

* Serious chronic disease (i.e., cardiac, renal, neurologic, metabolic, rheumatologic, psychiatric etc).
* Known or suspected impairment of immunologic function.
* Acute medical illness with or without fever within the last 72 hours or an oral temperature ≥ 100.4ºF (≥ 38.0ºC) at the time of inclusion.
* For the Menactra® and Menomune® groups, history of documented invasive meningococcal disease or previous meningococcal vaccination with the exception of meningococcal vaccination given as part of MTA02 trial.
* For the Control group, history of documented invasive meningococcal disease or previous meningococcal vaccination.
* Administration of immune globulin, other blood products within the last three months, injected or oral corticosteroids or other immunomodulatory therapy within six weeks of the study vaccine. Individuals on a tapering dose schedule of oral steroids lasting < 7 days may be included in the trial as long as they have not received more than one course within the last two weeks prior to enrollment.
* Antibiotic therapy within the 72 hours prior to vaccination or antibiotic therapy within the 72 hours prior to having any blood sample drawn.
* Received any vaccine in the 14-day period prior to study vaccination, or scheduled to receive any vaccination during the 14-day period after study vaccination.
* Suspected or known hypersensitivity to any of the vaccine components.
* Unavailable for the entire study period or unable to attend the scheduled visits or to comply with the study procedures.
* In females, a positive or equivocal urine pregnancy test at the time of vaccination.
* Enrolled in another clinical trial.
* Any condition, which, in the opinion of the investigator, would pose a health risk to the participant, or interfere with the evaluation of the vaccine.

Ages: 13 Years to 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 241 (Actual)
Dates: Start 2004-02; Primary Completion 2004-04 (Actual); Study Completion 2005-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Sanofi Pasteur Inc.
Locations (9):
- United States (9):
  - Atlanta, Georgia
  - Marietta, Georgia
  - Woburn, Massachusetts
  - Albany, New York
  - Akron, Ohio
  - Columbus, Ohio
  - Sellersville, Pennsylvania
  - Kingsport, Tennessee
  - Norfolk, Virginia

REFERENCES:
- [Result] Keyserling H, Papa T, Koranyi K, Ryall R, Bassily E, Bybel MJ, Sullivan K, Gilmet G, Reinhardt A. Safety, immunogenicity, and immune memory of a novel meningococcal (groups A, C, Y, and W-135) polysaccharide diphtheria toxoid conjugate vaccine (MCV-4) in healthy adolescents. Arch Pediatr Adolesc Med. 2005 Oct;159(10):907-13. doi: 10.1001/archpedi.159.10.907. PMID 16203934
- See also: Related Info — http://www.sanofipasteur.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited from 20 February 2004 to 08 April 2004 at 9 medical clinics in the US.
Pre-assignment Details: A total of 241 subjects that met the inclusion criteria were enrolled and vaccinated.
Groups:
- Menactra® Group: Subjects that received Menactra® vaccine in Study MTA02
- Menomune® Group: Subjects that received Menomune® vaccine in Study MTA02
- Control Group: Meningococcal vaccine-naïve subjects
Period: Overall Study
Arm/Group | Menactra® Group | Menomune® Group | Control Group
Started | 76 | 77 | 88
Completed | 76 | 77 | 88
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Menactra® Group | Menomune® Group | Control Group | Total
Number analyzed (Participants) | 76 | 77 | 88 | 241
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 56 | 57 | 68 | 181
  Between 18 and 65 years | 20 | 20 | 20 | 60
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 16.6 (1.91) | 16.8 (1.85) | 15.7 (1.97) | 16.4 (1.97)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 30 | 31 | 44 | 105
  Male | 46 | 46 | 44 | 136
Region of Enrollment [Number; unit: participants]
  United States | 76 | 77 | 88 | 241

OUTCOME MEASURES:

1. Primary Outcome: Geometric Mean Titers (GMTs) of Serum Bactericidal Activity for Each of the 4 Vaccine Serogroups.
Description: Geometric mean titers and their 95% confidence interval of serum bactericidal activity for the 4 vaccine serogroups before vaccination, at 8 days post- and 28 days post-booster dose of Menactra vaccine or a primary dose of Menactra vaccine in the meningococcal vaccine-naïve Control group.
Time Frame: Day 0 and 8 and 28 days post-vaccination
Population: GMT results were on the per-protocol population for immunogenicity.
Measure: Geometric Mean (95% Confidence Interval); unit: Titer
Arm/Group | Menactra® Group | Menomune® Group | Control Group
Number analyzed (Participants) | 71 | 72 | 84
Titer
  Serogroup A (Day 0) | 1075.2 [763.6 to 1514.1] | 193.6 [113.7 to 329.9] | 83.3 [47.3 to 146.8]
  Serogroup A (Day 8) | 9300.5 [7539.3 to 11473.2] | 4423.9 [3272.7 to 5980.0] | 12897.1 [9908.1 to 16787.9]
  Serogroup A (Day 28) | 4300.9 [3408.5 to 5427.0] | 3219.9 [2413.6 to 4295.5] | 6239.2 [4922.7 to 7907.8]
  Serogroup C (Day 0) | 246.2 [139.2 to 435.5] | 124.4 [65.9 to 234.8] | 39.7 [24.1 to 65.2]
  Serogroup C (Day 8) | 17888.7 [14004.2 to 22850.7] | 1149.4 [692.8 to 1907.0] | 7003.3 [4979.4 to 9849.7]
  Serogroup C (Day 28) | 8601.8 [6552.2 to 11292.6] | 664.0 [396.3 to 1112.5] | 2802.3 [1932.3 to 4063.9]
  Serogroup Y (Day 0) | 570.0 [353.9 to 918.3] | 398.6 [259.8 to 611.7] | 204.3 [131.4 to 317.8]
  Serogroup Y (Day 8) | 13088.9 [9486.0 to 18060.2] | 3098.2 [2170.0 to 4423.4] | 7061.3 [5029.8 to 9913.2]
  Serogroup Y (Day 28) | 5821.0 [4140.6 to 8183.3] | 2489.6 [1786.5 to 3469.3] | 4411.8 [3117.8 to 6242.7]
  Serogroup W-135 (Day 0) | 451.0 [300.2 to 677.4] | 126.8 [80.0 to 200.9] | 23.0 [15.7 to 33.7]
  Serogroup W-135 (Day 8) | 9861.6 [7442.9 to 13066.4] | 2008.9 [1516.2 to 2661.9] | 6036.6 [4555.5 to 7999.3]
  Serogroup W-135 (Day 28) | 4882.9 [3712.1 to 6422.9] | 1625.5 [1250.6 to 2112.8] | 3018.3 [2369.7 to 3844.4]

ADVERSE EVENTS:
Time Frame: Adverse events data were collected from the day of vaccination for 28 days post-vaccination.
Arm/Group | Menactra® Group | Menomune® Group | Control Group
Serious Adverse Events (participants affected / at risk) | 0/76 | 0/77 | 0/88
Other Adverse Events (participants affected / at risk) | 7/76 | 5/77 | 9/88
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Menactra® Group (N=76) | Menomune® Group (N=77) | Control Group (N=88)
Dysmenorrhoea (Reproductive system and breast disorders) | 1 (1) | 3 (3) | 5 (5)
Pharyngolaryngeal pain (Respiratory, thoracic and mediastinal disorders) | 6 (6) | 2 (3) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor must have the opportunity to review at least 60 days prior to submission for publication or presentation. If review indicates that potentially patentable subject matter would be disclosed, publication or public disclosure may be delayed for a maximum of an additional 60 days to allow for filing the necessary patent applications.